CLINICAL TRIAL: NCT07153224
Title: Mentorship, Intraoperative Consultation, and Coaching for Resilience and Outcomes in Early-career Surgeons Through Collaborative Peer Environment (MICROSCOPE): a Prospective International Time-bound Project
Brief Title: The MICROSCOPE Project
Acronym: MICROSCOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M1
Record Dates: First submitted 2025-08-11; First posted 2025-09-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Early Career Surgeons; Mental Wellbeing; Patients Outcomes; Mentorship; Surgical Coaching; Intra-operative Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early-career surgeons: Early career surgeons mental wellbeing status in terms of burnout, resilience and perceived quality of life will be observed exploring the relationship with the peri-operative support measure received (mentorship, intraoperative consultation, surgical coaching or standard practice). Also the outcomes of patients operated on by early career surgeons will be studied. Furthermore potential relationship between perio-operative supporto measures, mental status and outcomes will be explored.
  Interventions: Behavioral: Peri-operative support measures [mentorship, intraoperative consult, surgical coaching, standard practice (no structured support)]

INTERVENTIONS:
Behavioral: Peri-operative support measures [mentorship, intraoperative consult, surgical coaching, standard practice (no structured support)] — Mentorship: Formal (assigned by an institution or via an official program) or informal (personal relationship built during the career pathway) professional guidance relationships that support early-career surgeons in clinical decision-making, technical development, and emotional processing.
  Surgical Coaching: Structured, feedback-oriented discussions or sessions aimed at performance enhancement and reflective practice Intraoperative Consultation (IOC): Real-time assistance or second opinions provided by a more experienced surgeon or peers during a surgical procedure Standard practice: the surgeon performs the procedure supported by one or multiple assistants, as per internal hospital protocols and national/local regulations, receiving and providing natural feedback without a structured support system.

SUMMARY:
This multicenter observational prospective study aims to explore the impact of peri-operative support measures (mentorship or coaching or intraoperative consultation) on the mental well-being of early career surgeons. Furthermore sub-analyses will be conducted to explore the impact that surgeons mental wellbeing related to different support measures could have on patients' outcomes

DETAILED DESCRIPTION:
The MICROSCOPE study is a prospective, international, observational project evaluating the impact of structured perioperative support-mentorship, intraoperative consultation (IOC), and surgical coaching-on the well-being of early-career surgeons and their patients' outcomes.

Early-career surgeons (within 10 years post-training) face high stress, with limited structured support. This study investigates whether professional guidance improves surgeon resilience, reduces burnout, and enhances performance.

The project includes two components:

Surgeon-level study: Participants are observed over 12 months and grouped by support type received. Mental health outcomes are assessed using validated tools (Maslach Burnout Inventory, CD-RISC-10, QoL scale), alongside self- and assistant-rated performance metrics.

Patient-level study: Adult patients operated on by enrolled surgeons during the first 3 months are followed for 90 days. Outcomes include postoperative complications (CCI®, Clavien-Dindo), intraoperative events (Satava), reoperation, readmission, and mortality.

Data are collected via REDCap and analyzed using adjusted mixed-effects models to account for clustering and confounders. The study is investigator-initiated, with no external funding, and adheres to ethical standards including local IRB approval and informed consent.

MICROSCOPE aims to generate real-world evidence on how structured support can improve both surgical care quality and surgeon well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) treated for abdominal general surgical conditions in the emergency or elective setting or for thoraco-abdominal traumatic diseases. The list of surgical procedures is reported in the Supplementary Material 1
* Surgeries performed in elective, trauma, or emergency general surgery care

Exclusion Criteria:

* Patients operated by surgeons who completed general surgery residency more than 10 years before the study start date
* Pediatric patients < 18 years of age
* Patients or surgeons not willing to give their consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early career surgeons: graduating in general surgery in the last 10 years Surgeons performing elective general surgery, emergency general surgery and trauma surgery
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Burnout: Emotional Exhaustion | Baseline, Perioperative, 3 months, 6 months
  Maximun score 48. High scores relate to higher Emotional Exhaustion, contributing to higher burnout

SECONDARY OUTCOMES:
Burnout: Depersonalization | Baseline, Perioperative, 3 months, 6 months
  Depersonalizzation (DP) considering the treshold of 10 points from the Maslach Burnout Inventory
Psychological resilience | Baseline, Perioperative, 3 months, and 6 months
  Maximum score 40. High scores relate to higher resilience, contributing to potentially higher well-being
Perceived Surgical Performance | Perioperative
  Sefl evaluation by the surgeon using a 5-point Likert scale (1) a procedure that did not go well at all, (2) a procedure that could have gone better, (3) a regular procedure, (4) a successful procedure, (5) a highly successful procedure
Perceived Surgical Performance by the assistant | Perioperative
  Evaluation by the assistant using a 5-point Likert scale (1) a procedure that did not go well at all, (2) a procedure that could have gone better, (3) a regular procedure, (4) a successful procedure, (5) a highly successful procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Piero Bernardo Cioffi, MD, Principal Investigator — Niguarda Hospital
Locations (1):
- ASST GOM Niguarda, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The MICROSCOPE project is committed to ensuring reproducibility and transparency in its research practices. To support this, the following measures will be implemented:
  The study protocol and statistical analysis plan (SAP) will be registered and publicly available on Clinicaltrials.gov upon study initiation.
  Core study instruments will be documented and shared as supplementary materials in publications where possible.
  Statistical code used for primary and secondary outcome analyses will be made available upon reasonable request, subject to data-sharing agreements and institutional approvals.
  Deidentified, aggregate-level data may be shared with external collaborators for secondary analysis, conditional on ethical approval and collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After data collection completion, at least 12 months after study start date and for 1 year after then.
Access Criteria: Upon reasonable request to the study principal investigator